CLINICAL TRIAL: NCT05289297
Title: Karydakis Flap Procedure Versus Burow's Triangle Advancement Flap Procedure in the Surgical Treatment of Sacrococcygeal Pilonidal Sinus Disease
Brief Title: Karydakis Flap Versus Burow's Triangle Advancement Flap in the Surgery of Sacrococcygeal Pilonidal Sinus Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Sultanbeyli State Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022s01
Record Dates: First submitted 2022-03-13; First posted 2022-03-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pilonidal Sinus; Sacrococcygeal Pilonidal Disease
Keywords: Karydakis Flap; Pilonidal Cyst
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Karydakis Flap Procedure (Active Comparator): Vertical eccentric elliptical incision down to the post-sacral fascia, complete removal of unhealthy tissue, and normal tissue around the cyst and sinus tracts. Mobilization of the medial wound edge and advancement of the skin. Flap along the midline to the post-sacral fascia and suturing its margin to the lateral wound margin.
  Interventions: Procedure: Karydakis Flap Procedure
- Burow's Triangle Advancement Flap Procedure (Active Comparator): The flap is incised along the base of the wedge-shaped defect, and a small Burow's triangle is excised on the opposite side. The skin is mobilized and shifted in the direction of the arrow to close the defect. Excising the small Burow's triangle eliminates a dog ear at the base of the flap.
  Interventions: Procedure: Burow's Triangle Advancement Flap Procedure

INTERVENTIONS:
Procedure: Karydakis Flap Procedure — Pilonidal sinus surgery will be performed with the Karydakis Flap procedure.
  Arms: Karydakis Flap Procedure
Procedure: Burow's Triangle Advancement Flap Procedure — Pilonidal sinus surgery will be performed with the Burow's Triangle Advancement Flap procedure.
  Arms: Burow's Triangle Advancement Flap Procedure

SUMMARY:
In this study, we aim to compare the Karydakis flap and Burow's Triangle Advancement Flap techniques applied in the surgical treatment of pilonidal sinus in terms of complications, time to return to normal activity, and recurrence.

DETAILED DESCRIPTION:
Pilonidal sinus disease (PSD) is a chronic and inflammatory disease that is often generated in the sacrococcygeal region. It is commonly observed in puberty and young adult period and usually affects men. The incidence of pilonidal sinus disease is 26:100,000 and rising globally.

PSD risk factors contain young age, obesity, male gender, Mediterranean ethnicity, deep natal cleft, hairiness, and poor hygiene. It has been shown that PSD incidence increases in parallel with body weight. The precise etiology of pilonidal sinus disease is unclear. Many conservative and surgical methods have been described in treating pilonidal sinus disease. After the sinus area is excised, excision with laying open (secondary healing), excision with primary closure, marsupialization, and various flap techniques can be applied in surgical treatment. The primary principle in treatment is to ensure that the patient returns to normal life as soon as possible and eliminate recurrences. Although the best surgical technique in treating pilonidal sinus is controversial, the ideal operation should be cost-effective, simple to perform, short hospital stay, and have a low recurrence and complication rates. There is no definite consensus on an ideal technique yet.

In this study, we aim to compare the Karydakis flap and Burow's Triangle Advancement Flap techniques applied in the surgical treatment of pilonidal sinus in our clinic in terms of complications (wound dehiscence, seroma, hematoma, surgical site infection), time to return to normal activity, and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65
* Primary pilonidal sinus disease
* No abscess and absence of active infection during the operation

Exclusion Criteria:

* Patients under the age of 18 and over the age of 65
* Recurrent pilonidal sinus cases
* Patients with chronic comorbidities such as immunosuppression, collagen tissue disease, insulin-dependent diabetes mellitus, and neurological disease
* Patients with an ASA score of 3-4
* Patients with a body mass index greater than 35 kg/m2
* Patients with drug and alcohol addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-12 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain score according to the visual analogue scale | 1-3 days
  Postoperative pain after surgery ( measured by the visual analog score with 1 being minimum score and 10 being maximum score)
Postoperative wound healing time | 4 to 6 weeks
  Number of weeks of complete duration epithelialization of the wound
Procedure-related complications | 1 to 6 weeks
  Number of complications; related to the surgery, Type (wound dehiscence, seroma, hematoma, surgical site infection)
Time to return to normal activity | 4 to 6 weeks
  The number of weeks it passes the patient to return to normal activity.

SECONDARY OUTCOMES:
Recurrence of Pilonidal Sinus | 6 - 12 months
  Number of patients with recurrence pilonidal disease

CONTACTS AND LOCATIONS:
Overall Officials: Muhammer Ergenç, MD, Principal Investigator — Istanbul Sultanbeyli State Hospital
Locations (1):
- Istanbul Sultanbeyli State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doll D, Orlik A, Maier K, Kauf P, Schmid M, Diekmann M, Vogt AP, Stauffer VK, Luedi MM. Impact of geography and surgical approach on recurrence in global pilonidal sinus disease. Sci Rep. 2019 Oct 22;9(1):15111. doi: 10.1038/s41598-019-51159-z. PMID 31641150
- [Background] Harries RL, Alqallaf A, Torkington J, Harding KG. Management of sacrococcygeal pilonidal sinus disease. Int Wound J. 2019 Apr;16(2):370-378. doi: 10.1111/iwj.13042. Epub 2018 Nov 15. PMID 30440104
- [Background] Luedi MM, Schober P, Stauffer VK, Diekmann M, Doll D. Global Gender Differences in Pilonidal Sinus Disease: A Random-Effects Meta-Analysis. World J Surg. 2020 Nov;44(11):3702-3709. doi: 10.1007/s00268-020-05702-z. Epub 2020 Jul 17. PMID 32681319
- [Background] Alvandipour M, Zamani MS, Ghorbani M, Charati JY, Karami MY. Comparison of Limberg Flap and Karydakis Flap Surgery for the Treatment of Patients With Pilonidal Sinus Disease: A Single-Blinded Parallel Randomized Study. Ann Coloproctol. 2019 Dec 31;35(6):313-318. doi: 10.3393/ac.2018.09.27. Epub 2019 May 22. PMID 31113167
- [Background] Can MF, Sevinc MM, Hancerliogullari O, Yilmaz M, Yagci G. Multicenter prospective randomized trial comparing modified Limberg flap transposition and Karydakis flap reconstruction in patients with sacrococcygeal pilonidal disease. Am J Surg. 2010 Sep;200(3):318-27. doi: 10.1016/j.amjsurg.2009.08.042. Epub 2010 Feb 1. PMID 20122682
- [Background] Arslan K, Said Kokcam S, Koksal H, Turan E, Atay A, Dogru O. Which flap method should be preferred for the treatment of pilonidal sinus? A prospective randomized study. Tech Coloproctol. 2014 Jan;18(1):29-37. doi: 10.1007/s10151-013-0982-2. Epub 2013 Feb 21. PMID 23430349
- [Background] Oberemok S, Eliezri Y, Desciak E. Burow's wedge flap revisited. Dermatol Surg. 2005 Feb;31(2):210-6; discussion 216. doi: 10.1111/j.1524-4725.2005.31043. No abstract available. PMID 15762217
- [Background] Bali I, Aziret M, Sozen S, Emir S, Erdem H, Cetinkunar S, Irkorucu O. Effectiveness of Limberg and Karydakis flap in recurrent pilonidal sinus disease. Clinics (Sao Paulo). 2015 May;70(5):350-5. doi: 10.6061/clinics/2015(05)08. Epub 2015 May 1. PMID 26039952
- [Background] Ergenç, M., Uprak, T.K. Gender-specific prevalence of sacrococcygeal pilonidal sinus disease in Turkey: A retrospective analysis of a large cohort. Eur Surg 55, 43-47 (2023). https://doi.org/10.1007/s10353-022-00777-5